CLINICAL TRIAL: NCT03816878
Title: An Exploration of a Prime-Boost Approach for Universal Influenza Vaccination: Immunogenicity and Safety Study of Inactivated Subunit H5N1 Influenza Vaccine in Prior Recipients of Live Attenuated H2N2, H6N1 and H9N2 Influenza Vaccines and in H5N1 and Live Attenuated Vaccine Naïve Individuals
Brief Title: Immunogenicity and Safety Study of Inactivated Subunit H5N1 Influenza Vaccine in Prior Recipients of Live Attenuated H2N2, H6N1 and H9N2 Influenza Vaccines and in H5N1 and Live Attenuated Vaccine Naïve Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIR 327
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: pLAIV Recipients (Experimental): Participants who have received the pandemic live attenuated influenza vaccines (pLAIVs) H2N2, H6N1, or H9N2 during a previous CIR study will receive a single dose of 0.5 mL H5N1 pISV vaccine at Day 0.
  Interventions: Biological: H5N1 pISV
- Cohort 2: pLAIV Naive (Experimental): Participants who have never previously received a pLAIV will receive one dose of 0.5 mL H5N1 pISV vaccine at Day 0.
  Interventions: Biological: H5N1 pISV

INTERVENTIONS:
Biological: H5N1 pISV — Administered as an intramuscular (IM) injection

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of inactivated subunit H5N1 influenza vaccine in individuals who have previously received live attenuated H2N2, H6N1, or H9N2 influenza vaccine, as well as in individuals who have never previously received H5N1 or other pandemic live attenuated influenza vaccines.

DETAILED DESCRIPTION:
This study will evaluate the immunogenicity and safety of inactivated subunit H5N1 influenza vaccine in individuals who have previously received live attenuated H2N2, H6N1, or H9N2 influenza vaccine, as well as in individuals who have never previously received H5N1 or other pandemic live attenuated influenza vaccines (pLAIVs).

Participants will be enrolled in two cohorts. Cohort 1 will include participants who received two doses of live attenuated H2N2, H6N1, or H9N2 influenza vaccine during a prior Center for Immunization Research (CIR) study; Cohort 2 will include participants who have never previously received a pLAIV. Participants in both cohorts will receive one dose of H5N1 pISV vaccine by injection at Day 0.

Participants will attend study visits on Days 0, 7, 14, 28, 56, 90, and 360. Study visits may include a physical examination, medical history, and blood and urine collection. All participants will be followed for approximately 360 days after receiving the H5N1 pISV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 years and 60 years of age inclusive.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Available for the duration of the trial.
* Able to demonstrate understanding of key study concepts, study rationale, and study participation requirements by scoring greater than or equal to 70% on a written comprehension assessment in 3 or fewer attempts.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Willingness to allow storage and testing of laboratory samples for future research.
* Received 2 doses of live attenuated H2N2, H6N1, or H9N2 vaccine in a prior trial (Cohort 1) or H2N2, H6N1 and H9N2 naïve (Cohort 2)
* Willingness to forego seasonal influenza virus vaccination from 1 month before vaccination until 3 months after vaccination.
* Female subjects of childbearing potential must agree to have used effective birth control methods beginning at least one month prior to vaccination, and continuing with 'per label/fully effective use' for the chosen method for duration of the study, from amongst these:

  * pharmacologic/hormonal contraceptives, including oral, parenteral, subcutaneous, and transcutaneous delivery;
  * condoms with spermicide;
  * diaphragm with spermicide;
  * intrauterine device;
  * absolute abstinence from heterosexual intercourse as a matter of normal preferred lifestyle;
  * or must be surgically sterile or must be age 50 AND have had no menses at all for at least one full year.
  * All females must provide urine for pregnancy testing prior to enrollment (immediately prior vaccination), as well as a statement of menstrual history and a summary of all potentially reproductive sexual activity for the month prior to vaccination, and at each study contact throughout the study, and report known or suspected pregnancy immediately.
* Willingness to refrain from blood donation during the course of the study.

Exclusion Criteria:

* Pregnancy as determined by a positive test for human choriogonadotropin (beta-HCG), an indicator of pregnancy or history of recent unprotected intercourse in a woman of reproductive capacity.
* Currently breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hematologic, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Have medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* History of anaphylaxis in response to any vaccine or vaccine component.
* History of life-threatening reaction to prior influenza vaccine.
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory test for human immunodeficiency virus type 1 (HIV-1).
* Positive ELISA and confirmatory test (e.g., HCV RNA PCR) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome or history suggestive of impaired immune function.
* History of Guillain-Barré syndrome.
* Use of chronic oral or intravenous administration (greater than or equal to 14 days) of immunosuppressive doses of steroids, i.e., prednisone greater than 10 mg per day, immunosuppressants or other immune-modifying drugs within 30 days of starting this study.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study vaccination.
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study vaccination.
* Receipt of another investigational vaccine or drug within 30 days prior to study vaccination.
* In addition to the above, participants in Cohort 1 (pandemic live attenuated influenza vaccine [pLAIV] recipients) and Cohort 2 (naïve cohort) must also not experience any of the following:

  * Previous enrollment in an H5N1 influenza vaccine trial.
* Participants in Cohort 2 (naïve cohort) will be excluded if they are:

  * Seropositive to the H5N1 influenza A virus (serum hemagglutination inhibition assay (HAI) titer greater than 1:8).
  * Have previously received an investigational live attenuated influenza vaccine (LAIV) in another study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R. Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: pLAIV Recipients | Cohort 2: pLAIV Naive
Started | 11 | 21
Completed | 10 | 20
Not Completed | 1 | 1
Not completed — Taken off study after Day 28 due to unrelated serious adverse event requiring hospitalization | 1 | 0
Not completed — Volunteer taken off study due to incarceration | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: pLAIV Recipients | Cohort 2: pLAIV Naive | Total
Number analyzed (Participants) | 11 | 20 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 20 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.7 [36 to 58] | 38 [27 to 58] | 41 [27 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 4 | 14 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 10 | 19 | 29
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 20 | 31

OUTCOME MEASURES:

1. Primary Outcome: Fold Rise in Titer of Anti-group 1 Stalk-antibodies in Recipients of the Pandemic Live Attenuated Influenza Vaccines (pLAIVs) (H2N2, H6N1 and H9N2) Compared to the Control pLAIV-naïve Cohort
Description: As measured by enzyme-linked immunosorbent assay (ELISA) and microneutralization assay (MN) using the chimeric cH6/N1 probe
Time Frame: Measured through Day 28
Measure: Geometric Mean (Standard Deviation); unit: fold rise
Arm/Group | Cohort 1: pLAIV Recipients | Cohort 2: pLAIV Naive
Number analyzed (Participants) | 11 | 20
fold rise
  Day 0 | 1.5 (1.2) | 1 (0)
  Day 28 | 1.4 (1.2) | 1 (0)

2. Secondary Outcome: Number of Participants With Vaccine-related Adverse Events in the pLAIV Compared to the Control Cohort
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Time Frame: Measured through Day 28 for non serious adverse events
Measure: Number; unit: number of participants
Arm/Group | Cohort 1: pLAIV Recipients | Cohort 2: pLAIV Naive
Number analyzed (Participants) | 11 | 20
number of participants
  Injection site erythema | 0 | 1
  Injection site induration | 1 | 0
  Injection site pain | 1 | 5
  Malaise | 1 | 1
  Pain | 1 | 0

ADVERSE EVENTS:
Time Frame: 90 days beginning at study vaccination
Arm/Group | Cohort 1: pLAIV Recipients | Cohort 2: pLAIV Naive
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/20
Other Adverse Events (participants affected / at risk) | 8/11 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: pLAIV Recipients (N=11) | Cohort 2: pLAIV Naive (N=20)
Surgery (Gastrointestinal disorders) | 1 (1) | NA (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: pLAIV Recipients (N=11) | Cohort 2: pLAIV Naive (N=20)
Blood pressure increased (Cardiac disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth Disorder (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 5 (5)
Malaise (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT03816878/Prot_SAP_001.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03816878/ICF_000.pdf